CLINICAL TRIAL: NCT07347808
Title: A Phase 1, Single-Dose, Open-Label, Parallel-Group Pharmacokinetic Study of VCT220 in Subjects With Moderate Renal Impairment and Matched Subjects With Normal Renal Function
Brief Title: A Pharmacokinetic Study of VCT220 With Moderate Renal Impairment Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vincentage Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VCT220-I-08
Record Dates: First submitted 2025-12-22; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Subjects with Moderate Renal Impairment (absolute eGFR ≥30 and <60 mL/min)
  Interventions: Drug: VCT220
- Group B (Experimental): Subjects with Normal Renal Function Matched to Subjects with Moderate Renal Impairment (absolute eGFR ≥90 and <130 mL/min)
  Interventions: Drug: VCT220

INTERVENTIONS:
Drug: VCT220 — Single oral dose of VCT220 40 mg administered after a standardized breakfast.

SUMMARY:
This Phase 1 study is designed to evaluate the pharmacokinetics and safety of a single oral dose of VCT220 (other name: CX11) in subjects with moderate renal impairment compared with age-, sex-, and body mass index (BMI)-matched subjects with normal renal function. The results of this study will provide scientific evidence to support appropriate clinical dosing recommendations of VCT220 in subjects with renal impairment.

DETAILED DESCRIPTION:
This is a single-center, single-dose, open-label, non-randomized, parallel-group Phase 1 study. Subjects with moderate renal impairment (absolute estimated glomerular filtration rate [eGFR] ≥30 and <60 mL/min) and matched subjects with normal renal function (absolute eGFR ≥90 and <130 mL/min) will be enrolled.

Subjects will receive a single oral dose of VCT220 40 mg following a standardized breakfast. Pharmacokinetic blood samples will be collected up to 72 hours post-dose to characterize the plasma pharmacokinetics of VCT220 and its metabolite VCT289. Safety will be assessed through monitoring of adverse events, vital signs, physical examinations, laboratory tests, and electrocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 75 years
* Body mass index (BMI) between 18.5 and 32.0 kg/m²
* Able and willing to provide written informed consent
* Willing to comply with contraception requirements
* Moderate renal impairment group
* Absolute eGFR ≥30 and <60 mL/min
* Diagnosis of chronic kidney disease for ≥3 months with stable renal function
* Normal renal function group:

Absolute eGFR ≥90 and <130 mL/min Matched to moderate renal impairment subjects by sex, age (±10 years), and BMI (±10%)

Exclusion Criteria:

* History of hypersensitivity to GLP-1 receptor agonists or study drug components
* History of hypoglycemia
* History or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2
* History of pancreatitis
* Clinically significant cardiovascular, hepatic, gastrointestinal, neurological, hematologic, endocrine, or psychiatric disease
* Use of prohibited medications affecting drug metabolism prior to dosing
* Positive tests for hepatitis B, hepatitis C, HIV, or syphilis
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-03-13 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of VCT220 | Day 1 at 0 h prior to dosing and at 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, and 24.0 h (Day 2) ,36.0 h(Day 2) , 48.0 h (Day 3), and 72.0 h (Day 4) after dosing
Area Under the Plasma Concentration-Time Curve From Time 0 to Last Measurable Concentration (AUC₀-t) of VCT220 | Day 1 at 0 h prior to dosing and at 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, and 24.0 h (Day 2) ,36.0 h(Day 2) , 48.0 h (Day 3), and 72.0 h (Day 4) after dosing

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From dosing through safety follow-up (Day 7 ± 3 days)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No